CLINICAL TRIAL: NCT06383091
Title: Impact of Manual Therapy on Laryngeal Function Following Total Thyroidectomy
Acronym: Man Total Thy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00380938
Record Dates: First submitted 2024-04-15; First posted 2024-04-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Total Thyroidectomy
Keywords: manual; pain neuroscience education; total thyroidectomy; Speech Pathology

STUDY DESIGN:
Intervention Model Description: This is meant to be a parallel study. However, The Speech Language Pathologists will not be blinded as the Speech Pathologists are providing each regimen. If a participant in either group requires more intensive sessions or a differing regimen given the severity of complaints, the participants will receive it as per the recommendation of the Speech-Language Pathologist so as not to unblind the PI. An intent to treat analysis will be performed to accurately describe the data in the case of crossover and/or dropout.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck Manual, Stretches, Pain Neuroscience Education with Voice Exercise and Scar Massage Arm (Active Comparator): Patients will receive direct manual massage to the anterior neck, general neck stretches and pain neuroscience education along with voice exercises and scar massage with a trained Speech-Language Pathologist
  Interventions: Behavioral: Anterior Neck Manual Therapy; Behavioral: Pain Neuroscience Education; Behavioral: Neck Stretches; Behavioral: Scar massage; Behavioral: Voice Exercises
- Voice Exercises and Scar Massage with placebo Manual/Stretching and Pain Education (Placebo Comparator): Patients will be given voice exercise and scar massages with a trained Speech Language Pathologist, alongside placebo manual/stretching and placebo pain education.
  Interventions: Behavioral: Scar massage; Behavioral: Voice Exercises; Behavioral: Placebo Anterior Neck Manual Therapy; Behavioral: Placebo Pain Neuroscience Education; Behavioral: Placebo Neck Stretches

INTERVENTIONS:
Behavioral: Anterior Neck Manual Therapy — Manual massage applied to the anterior neck, including hyolaryngeal elevators, depressors, sternocleidomastoid.
  Arms: Neck Manual, Stretches, Pain Neuroscience Education with Voice Exercise and Scar Massage Arm
Behavioral: Pain Neuroscience Education — Description of how the pain system works from a neurobiological level, discussing the biopsychosocial model that influences pain.
  Arms: Neck Manual, Stretches, Pain Neuroscience Education with Voice Exercise and Scar Massage Arm
Behavioral: Neck Stretches — Bilateral cervical side bending, cervical extension and bilateral rotational neck stretches held for 20 seconds x3.
  Arms: Neck Manual, Stretches, Pain Neuroscience Education with Voice Exercise and Scar Massage Arm
Behavioral: Scar massage — Digital manipulation of the scar itself in circles.
Behavioral: Voice Exercises — Stemple Voice Exercises
Behavioral: Placebo Anterior Neck Manual Therapy — Will apply extremely light manual contact to the anterior neck, including hyolaryngeal elevators, depressors, sternocleidomastoid.
  Arms: Voice Exercises and Scar Massage with placebo Manual/Stretching and Pain Education
Behavioral: Placebo Pain Neuroscience Education — Will discuss how pain will as a result of the surgical intervention.
  Arms: Voice Exercises and Scar Massage with placebo Manual/Stretching and Pain Education
Behavioral: Placebo Neck Stretches — Will ask patient to look down as a neck stretch held for 20 seconds x3.
  Arms: Voice Exercises and Scar Massage with placebo Manual/Stretching and Pain Education

SUMMARY:
In this clinical trial, the investigators are seeking to learn if a course of voice therapy, including neck massage, stretches and pain science education in addition to voice exercise and scar massage will effectively treatment patient complaints of swallowing or voice changes after total thyroidectomy as compared to voice exercise and scar massage alone.

The main questions it aims to answer are:

Will neck massage, stretches and pain science education reduce patient complaints of swallowing changes after total thyroidectomy?

Will neck massage, stretches and pain science education reduce patient complaints of voice changes after total thyroidectomy?

Will neck massage, stretches and pain science education reduce patient complaints of scar tethering and quality changes after total thyroidectomy?

Will neck massage, stretches and pain science education improve quality of life after total thyroidectomy?

Participants will:

Participate in 4 visits with the participant's endocrine/laryngology surgeon. One prior and 3 after surgery for endoscopic evaluation and tests.

Participate in 5 Speech-Language Pathology Sessions for intervention exercises and tests. One prior and 4 after surgery.

Complete a journal of the participant's Home Exercise Practice

ELIGIBILITY:
Inclusion Criteria:

* The study population consists of individuals with malignant or benign thyroid disease scheduled to undergo total thyroidectomy
* native speakers of English
* All patients will be greater than or equal to 18 years of age

Exclusion Criteria:

* Participants will be excluded if they have completed voice therapy prior
* are current smokers
* have organic vocal fold pathology or clear mucosal changes to the vocal folds that can affect vibration (e.g., vocal fold scar, polyp, or nodules),
* pre-existing unilateral or bilateral vocal fold paralysis
* have had prior surgical neck or chest history including central or lateral neck dissection
* pre- or post-operative abscess or inflammation
* have a history of radiation, chronic cervical pain or cervicalgia, abnormal baseline swallowing
* have underlying and, or plan to change supplemental hormones
* greater than 10% otherwise unexplained weight loss
* had a recent aspiration pneumonia
* history of esophageal interventions or surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Acoustic measures of voice clarity | Baseline, 1 year
  Acoustic measurement of relative Cepstral Peak Prominence (dB) in a speaking voice sample.
Acoustic measures of speaking voice pitch | Baseline, 1 year
  Acoustic measurement of average fundamental speaking pitch in Hertz before and after surgery.
Acoustic measures of speaking voice quality subjectively | Baseline, 1 year
  Clinicians will rate each patient's voice as having or not having each of the following perceptual qualities: Grade, Roughness, Asthenia, Breathiness, Strain. The scale is as follows: 0 (no perceptual quality) to 3 (severe perceptual quality).
Swallowing Quality of Life as assessed by the Eating Assessment Tool - 10 | Baseline, 1 year
  Patients will rate themselves from a 0 - 4 (0: no problem to 4: Severe Problem) on 10 items within the Eating Assessment Tool - 10
Laryngeal sensation | Baseline, 1 year
  Using a visual analogue scale of pain - from 0: no pain, to 10: worst pain. Patients will rate their pain.
Scar Tethering Distance | Baseline, 1 year
  Distance in centimeters will be measured between the hyoid bone and scar with swallowing.
Scar Quality as assessed by The Patient and Observer Scar Assessment Scale | Baseline, 1 year
  The Patient and Observer Scar Assessment Scale will be used to measure from 0: normal skin, to 10: worst scar imaginable.
Voice Quality of Life as measures by the Voice Related Quality of Life - 10 | Baseline, 1 year
  Quality of life measures: On a raw scale from 10 - 50 : 10 being no impact on quality of life, and 50 being the greatest impact on quality of life, participants will rate themselves.

SECONDARY OUTCOMES:
Adverse Effects in the Experimental Group | Baseline, 1 year
  Will document the total number of adverse effects in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Vaninder Dhillon, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruno G, Melissa S, Natalia C, Francesco G, Francesco F, Rocco B, Patrizia L, Antonella P, Ettore C, Zhang D, Gianlorenzo D, Francesco G. Posture and dysphonia associations in patients undergoing total thyroidectomy: stabilometric analysis. Updates Surg. 2020 Dec;72(4):1143-1149. doi: 10.1007/s13304-020-00844-0. Epub 2020 Jul 11. PMID 32654042
- [Background] Lee JS, Kim JP, Ryu JS, Woo SH. Effect of wound massage on neck discomfort and voice changes after thyroidectomy. Surgery. 2018 Nov;164(5):965-971. doi: 10.1016/j.surg.2018.05.029. Epub 2018 Jul 24. PMID 30054014
- [Background] McMillan H, Barbon CEA, Cardoso R, Sedory A, Buoy S, Porsche C, Savage K, Mayo L, Hutcheson KA. Manual Therapy for Patients With Radiation-Associated Trismus After Head and Neck Cancer. JAMA Otolaryngol Head Neck Surg. 2022 May 1;148(5):418-425. doi: 10.1001/jamaoto.2022.0082. PMID 35297966
- [Background] Pattanshetty RB, Patil SN. Role of Manual Therapy for Neck Pain and Quality of Life in Head and Neck Cancer Survivors: A Systematic Review. Indian J Palliat Care. 2022 Jan-Mar;28(1):99-112. doi: 10.25259/IJPC_10_2021. Epub 2021 Dec 18. PMID 35673382
- [Background] Ribeiro VV, Pedrosa V, Silverio KCA, Behlau M. Laryngeal Manual Therapies for Behavioral Dysphonia: A Systematic Review and Meta-analysis. J Voice. 2018 Sep;32(5):553-563. doi: 10.1016/j.jvoice.2017.06.019. Epub 2017 Aug 26. PMID 28844806